CLINICAL TRIAL: NCT01562184
Title: A Controlled Trial of Transcranial Direct Current Stimulation as a Treatment for Unipolar and Bipolar Depression
Brief Title: Investigating tDCS as a Treatment for Unipolar and Bipolar Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Duke University (Other); Emory University (Other); Sheppard Pratt Health System (Other); University of Medicine and Dentistry of New Jersey (Other); University of Texas (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC11515; #11T-005 (Other Grant/Funding Number: Stanley Medical Research Institute)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Unipolar Depression; Bipolar Depression
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS (Active Comparator): Active tDCS
  Interventions: Device: Soterix tDCS device
- Sham tDCS (Sham Comparator): Sham tDCS
  Interventions: Device: Sham tDCS device

INTERVENTIONS:
Device: Sham tDCS device — Sham tDCS
  Arms: Sham tDCS
Device: Soterix tDCS device — Active tDCS
  Arms: Active tDCS

SUMMARY:
Transcranial direct current stimulation (tDCS) is a novel treatment approach for depression that has shown promising efficacy in four recent double-blind, randomized, sham-controlled trials (RCT) and a meta-analysis. This study is a RCT of tDCS in depressed patients, testing its efficacy in both unipolar and bipolar depression. Mood, cognitive test performance and biomarkers will be measured during the trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above.
* Meets criteria for a DSM-IV Major Depressive Episode with duration of at least 4 weeks.
* Total score ≥ 20 on the Montgomery-Asberg Depression Rating Scale at study entry.

Exclusion Criteria:

* Current episode duration greater than 3 years.
* Failed more than 3 adequate antidepressant trials in current episode.
* DSM-IV psychotic disorder.
* Drug or alcohol abuse or dependence (preceding 3 months).
* Inadequate response to ECT in the current episode of depression.
* Rapid clinical response required, e.g., high suicide risk.
* Significant acute suicide risk, defined as follows: suicide attempt within the previous 6 months that required medical treatment; or ≥ 2 suicide attempts in the past 12 months; or has a clear-cut plan for suicide and states that they cannot guarantee that they will call their regular psychiatrist or the investigator if the impulse to implement the plan becomes substantial during the study; or in the investigator's opinion, is likely to attempt suicide within the next 6 months.
* Clinically defined neurological disorder or insult.
* Metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
* Pregnancy.
* Concurrent long acting benzodiazepines, ritalin or dexamphetamine medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS) | 12 weeks

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR) | 12 weeks
Montreal Cognitive Assessment (MoCA): Global Cognitive Function | 8 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Emory University, Atlanta, Georgia
  - Sheppard Pratt, Towson, Maryland
  - Rowan University, Cherry Hill, New Jersey
  - Duke University, Durham, North Carolina
  - University of Texas Southwestern, Dallas, Texas
- University of New South Wales / Black Dog Institute, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Martin DM, McClintock SM, Aaronson ST, Alonzo A, Husain MM, Lisanby SH, McDonald WM, Mohan A, Nikolin S, O'Reardon J, Weickert CS, Loo CK. Pre-treatment attentional processing speed and antidepressant response to transcranial direct current stimulation: Results from an international randomized controlled trial. Brain Stimul. 2018 Nov-Dec;11(6):1282-1290. doi: 10.1016/j.brs.2018.08.011. Epub 2018 Aug 23. PMID 30172724
- [Derived] Loo CK, Husain MM, McDonald WM, Aaronson S, O'Reardon JP, Alonzo A, Weickert CS, Martin DM, McClintock SM, Mohan A, Lisanby SH; International Consortium of Research in tDCS (ICRT). International randomized-controlled trial of transcranial Direct Current Stimulation in depression. Brain Stimul. 2018 Jan-Feb;11(1):125-133. doi: 10.1016/j.brs.2017.10.011. Epub 2017 Oct 27. PMID 29111077